CLINICAL TRIAL: NCT02534792
Title: Early Revalvulation After Fallot Repair Improves Clinical Outcome
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S58389
Record Dates: First submitted 2015-08-25; First posted 2015-08-28 (Estimated); Last update posted 2016-10-27 (Estimated); Status verified 2016-10

CONDITIONS: Tetralogy of Fallot
MeSH Terms: conditions — Tetralogy of Fallot

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Revalvulation time early: Early revalvulation by homograft or percutaneous valve
  Interventions: Other: Revalvulation
- Revalvulation time late: Late revalvulation by homograft or percutaneous valve
  Interventions: Other: Revalvulation

INTERVENTIONS:
Other: Revalvulation

SUMMARY:
Aim With this retrospective study, the investigators would like to evaluate and, if possible confirm, whether earlier revalvulation of the right ventricular outflow tract is better than late revalvulation. Up to now, no analysis is done to validate this policy change.

Patient selection All patients registered in the database of paediatric and congenital cardiology of the University Hospitals in Leuven, with sufficient follow-up data, and who underwent transannular patching at repair will be included in the study.

Methodology and statistical analysis All files will be reviewed for demographic, electrocardiographic, echocardiographic, and outcome data. Besides descriptive statistics, Cox regression will be performed to detect whether the time period between repair and revalvulation influences clinical outcome (defined as death, heart failure hospitalization, redo-revalvulation, implantation of automatic defibrillator, endocarditis).

ELIGIBILITY:
Inclusion Criteria:

* Tetralogy of Fallot patients repaired with transannulaire patch.

Exclusion Criteria:

* None.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tetralogy of Fallot patients repaired with transannulaire patch.
Sampling Method: Non-Probability Sample
Enrollment: 320 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
death | 10 years

SECONDARY OUTCOMES:
endocarditis | 10 years
re-intervention | 10 years

CONTACTS AND LOCATIONS:
Locations (1):
- UZ Leuven, Leuven, Belgium